CLINICAL TRIAL: NCT04675047
Title: Multimodal Brain Decoding of Pain Sensitivity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM108044F
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy control: healthy control
  Interventions: Other: no intervention for healthy control

INTERVENTIONS:
Other: no intervention for healthy control — observational study - no intervention

SUMMARY:
Pain is the leading cause of disability worldwide. However, the pain sensitivity of individuals varies to a large extent, which often results in the mismatch between clinical diagnosis or treatment and individual's actual needs. There are still no established objective indicators for comparisons between individuals. This integrated pilot project is the first large-scale, multi-modal brain decoding study for pain sensitivity. We will explore the brain network signature of pain sensitivity by analyzing electroencephalogram (EEG) signals and magnetic resonance imaging (MRI.) Meanwhile, we will integrate the innate, environmental, and humanity factors with aforementioned brain network signatures to establish multi- modal objective model of pain sensitivity using machine learning. This research team is composed of more than 30 physicians, scientists, and IT experts, along with international collaborators with expertise in the fields of neuroscience, medical imaging, and human philosophy. The five elite groups constitute this international research team and establish five multi-disciplinary sub-projects: Sub-project A： Pain sensitivity and associated innate and environmental factors Sub-project B： Electrophysiological brain signatures of pain sensitivity Sub-project C： MRI brain signatures of pain sensitivity Sub-project D： Innovative brain computer interface (BCI) technology in pain sensitivity measurement and prediction Sub-project E： Pain and Art: neuro-mental mechanisms and potential applications There are three key features of this integrated project: scientific novelty, technology and humanity. In terms of scientific novelty, in addition to machine learning and big data applications, we will focus on the deep brain structure such as brainstem, in which the image acquisition has been difficult in the past. We will develop an MRI sequence and EEG protocol optimized for brainstem. In terms of technology, we will develop a wearable EEG cap implanted with algorithm chip for clinical measurement to decode the pain sensitivity real time. In terms of humanity, we will combine music and painting appreciation to explore their impact on brain signatures related to pain sensitivity. Furthermore, we will develop potential applications of art intervention in pain modulation. We expect this pilot project to achieve the four following goals:

1. To establish a Taiwan database of pain sensitivity. Meanwhile, to clarify the interactions between the innate and environmental factors of the individual and the brain network, and to identify brain signatures related to pain sensitivity. (sub- projects A, B, C)
2. To confirm the brain signatures for predicting the pain sensitivity using machine learning. In addition, to develop wearable devices such as EEG cap for large sample screening by combining the brain-computer interface through the industry-university cooperation (sub-projects B, C, D)
3. To explore the plasticity of brain signatures related to pain sensitivity by sensory modulation such as music, painting appreciation or transcutaneous electrical nerve stimulation, and to explore the application potential for pain modulation (sub-projects B, C, D, E)
4. Based on the cooperation model of this international research team, we will cultivate young researchers, and promote academic interactions among different team members, and improve the international visibility and competitiveness of Taiwan (sub-projects A, B, C, D, E)

ELIGIBILITY:
Inclusion Criteria:

* aged 20-55
* understand the study and provide informed consent

Exclusion Criteria:

* Any acute or chronic condition that could potentially affect pain perception, including diabetes, hypertension, peripheral and central nervous disorders
* Presence of any pain disorder or suffering from any acute pain within 2 weeks
* History of any neurological disease, except primary headache with headache frequency less than 1 days per month
* Psychiatric disorders including major depressive disorder, post-traumatic stress disorder, personality disorder, bipolar disorder, and schizophrenia
* History of substance abuse, including alcohol, analgesic, and illicit drugs.
* Any condition that would make participants contra-indicated to magnetic resonance imaging (MRI) scans transcutaneous electrical nerve stimulation (TENS), or electroencephalography (EEG).

Ages: 20 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Healthy control
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
sensory thresholds | 30 minutes
  Using quantitative sensory testing (QST) to evaluate the sensory threshold
EEG change (1) | 10 minutes
  Linear analysis of EEG with pain sensitivity
EEG change (2) | 10 minutes
  Nonlinear analysis of EEG with pain sensitivity
MRI | 90 minutes
  Analysis of MRI correlatin with pain sensitivity
fMRI | 90 minutes
  Analysis of fMRI correlatin with pain sensitivity
Humoral relationship (1) | 5 minutes
  Test the related hormones to evaluate the relationship with sensitivity
Humoral relationship (2) | 5 minutes
  Test the related cytokines to evaluate the relationship with sensitivity

SECONDARY OUTCOMES:
innate and environmental factors associated with pain sensitivity | 5 minutes
  explory potential factors that may influence the pain sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan